CLINICAL TRIAL: NCT02830243
Title: The Comparison of Analgesic Effect of Volatile Anesthetics Using Surgical Pleth Index
Brief Title: Comparison of Analgesic Effect of Volatile Anesthetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoungho Ryu, Clinical assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-05-058
Record Dates: First submitted 2016-07-09; First posted 2016-07-12 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Anesthesia was maintained with sevoflurane.
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Anesthesia was maintained with desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — End-tidal concentration of sevoflurane was maintained at age-corrected 1 minimum alveolar concentration throughout the study period. The remifentanil infusion rate was adjusted using TCI pump to achieve surgical pleth index between 20 and 50.
  Other Names: SEVO
  Arms: Sevoflurane
Drug: Desflurane — End-tidal concentration of desflurane was maintained at age-corrected 1 minimum alveolar concentration throughout the study period. The remifentanil infusion rate was adjusted using TCI pump to achieve surgical pleth index between 20 and 50.
  Other Names: DES
  Arms: Desflurane

SUMMARY:
The purpose of this clinical trial is to compare analgesic effect of sevoflurane and desflurane at equal minimum alveolar concentrations using surgical pleth index.

DETAILED DESCRIPTION:
Volatile anesthetics vary in their relative hypnotic potency. Recent studies demonstrated that equi-minimum alveolar concentration of various volatile anesthetic agents may produce different bispectral index values. However, the difference between analgesic effects of volatile anesthetics have not yet been investigated. The purpose of this clinical trial is to compare analgesic effect of sevoflurane and desflurane at equal minimum alveolar concentrations using surgical pleth index-guided remifentanil infusion.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing balanced general anesthesia using volatile anesthetics and remifentanil
* patients with american society of anesthesiologist physical status I, II
* patients aged 19-65 years
* patients obtaining written informed consent

Exclusion Criteria:

* patients with a history of any psychiatric or neurological disease
* patients who had received any medication affecting the central nervous system
* patients who had received medication affecting the sympathetic or parasympathetic nervous systems
* patients undergoing tracheal intubation for airway management
* pregnant women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-08 (Actual)

PRIMARY OUTCOMES:
Remifentanil consumption (µg/kg/min) | During the intraoperative period

SECONDARY OUTCOMES:
Target effective site concentration of remifentanil (ng/ml) | After at least 10 min of stable surgical pleth index values

CONTACTS AND LOCATIONS:
Overall Officials: Kyoungho Ryu, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ryu KH, Kim JA, Ko DC, Lee SH, Choi WJ. Desflurane reduces intraoperative remifentanil requirements more than sevoflurane: comparison using surgical pleth index-guided analgesia. Br J Anaesth. 2018 Nov;121(5):1115-1122. doi: 10.1016/j.bja.2018.05.064. Epub 2018 Jul 4. PMID 30336856